CLINICAL TRIAL: NCT00191191
Title: LY231514 500 mg/m2 and LY231514 1000 mg/m2 in Patients With Advanced Non-Small Cell Lung Cancer Who Were Previously Treated With Prior Systemic Anti Cancer Therapy: A Randomized Phase II Trial
Brief Title: To Investigate Efficacy and Safety of Pemetrexed as Second or Third Line Therapy in Patients With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5250; H3E-JE-NS01 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed 500 mg/m2 (Experimental): Pemetrexed 500 mg/m2
  Interventions: Drug: Pemetrexed 500 mg/m2
- Pemetrexed 1000 mg/m2 (Experimental): Pemetrexed 1000 mg/m2
  Interventions: Drug: Pemetrexed 1000 mg/m2

INTERVENTIONS:
Drug: Pemetrexed 500 mg/m2 — 500 mg/m2, intravenous (IV), every 21 days, one year from registration date
  Other Names: Alimta; LY231514
  Arms: Pemetrexed 500 mg/m2
Drug: Pemetrexed 1000 mg/m2 — 1000 mg/m2, intravenous (IV), every 21 days, one year from registration date
  Other Names: Alimta; LY231514
  Arms: Pemetrexed 1000 mg/m2

SUMMARY:
To investigate efficacy and safety of pemetrexed as second or third line therapy in patients with non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage III or IV
* Previously treated with one or two chemotherapeutic regimens
* Performance status: 0-2

Exclusion Criteria:

- Inability or unwillingness to take folic acid or vitamin B12 supplementation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time(UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gifu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline demographics and efficacy outcome measures are provided for the Full Analysis Set population (all randomized participants who met all inclusion and no exclusion criteria and received at least one dose of study drug).
Groups:
- Pemetrexed 500 mg/m2: Pemetrexed 500 mg/m2, intravenous, every 21 days
- Pemetrexed 1000 mg/m2: Pemetrexed 1000 mg/m2, intravenous, every 21 days
Period: Overall Study
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Started | 114 | 112
Safety Analysis Population | 114 | 111
Full Analysis Set Population | 108 | 108
Completed | 0 | 0
Not Completed | 114 | 112
Not completed — Entry Criteria Exclusion | 2 | 0
Not completed — Treated with Another Systemic Agent | 1 | 1
Not completed — Adverse Event | 11 | 21
Not completed — Progressive Disease | 84 | 72
Not completed — Toxicity After Dose Reduction | 7 | 8
Not completed — Family/Caregiver Decision | 5 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 2
Not completed — Good Clinical Practice Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2 | Total
Number analyzed (Participants) | 108 | 108 | 216
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.7) | 61.3 (8.8) | 61.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 68 | 69 | 137
Region of Enrollment [Number; unit: participants]
  Japan | 108 | 108 | 216
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 43 | 36 | 79
    1 - Ambulatory, Restricted Strenuous Activity | 59 | 66 | 125
    2 - Ambulatory, No Work Activities | 6 | 6 | 12
Histological Types [Number; unit: participants]
  Adenocarcinoma | 77 | 80 | 157
  Squamous Cell Carcinoma | 23 | 25 | 48
  Large Cell Carcinoma | 5 | 1 | 6
  Adenosquamous Carcinoma | 1 | 0 | 1
  Other | 2 | 2 | 4
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 161.0 (7.9) | 161.1 (8.7) | 161.0 (8.3)
Weight [Mean (Standard Deviation); unit: kilograms] | 59.8 (9.9) | 59.1 (11.9) | 59.5 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria as determined by the Case Judgment Committee. Best overall response was defined as the most favorable overall response recorded for each patient during the observation period. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 3.2 years)
Population: Full analysis set: all randomized participants who met all of the inclusion criteria and none of the exclusion criteria and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Number analyzed (Participants) | 108 | 108
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 20 | 16
  Stable Disease (SD) | 40 | 34
  Progressive Disease (PD) | 48 | 58

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression.
Time Frame: time of response to progressive disease (up to 3.2 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Number analyzed (Participants) | 108 | 108
months | 4.9 [3.8 to 8.7] | 3.0 [2.8 to 6.1]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from the scheduled date of the first treatment cycle until the date of confirmation of progressive disease on the overall response rating. For patients who died before confirmation of progressive disease, the number of days until the date of death (from any cause) was handled as progression-free survival.
Time Frame: baseline to measured progressive disease (up to 3.2 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Number analyzed (Participants) | 108 | 108
months | 3.0 [2.0 to 3.5] | 2.5 [1.8 to 3.2]

4. Secondary Outcome: Change From Baseline to 3 Months in Quality of Life Questionnaire for Cancer Patients Treated With Anticancer Drugs (QOL-ACD)
Description: 20-items assessed quality of life in patients undergoing chemotherapy. Scores range from 1 (not at all/very poor) to 5 (very much/very well). Face scale scores (patient circles number of the face that best fits his/her feelings) range from 1 (sad face) to 5 (smiling face). Item scores were grouped according to Functional (daily activity: 5 items), Physical (5 items), Emotional (psychological condition: 4 items), Social Attitude (5 items), and Face Scale (1 item). Score of subscales were converted to scores with range from 0 to 100. Higher scores represent higher QOL.
Time Frame: Baseline (pre-dose), 3 Months after first dose of Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Number analyzed (Participants) | 108 | 108
units on a scale
  Functional Baseline (n=107, n=107) | 77.0 (24.81) | 75.0 (26.18)
  Functional Change from Baseline (n=58, n=60) | -1.5 (23.66) | -3.7 (19.99)
  Physical Baseline (n=107, n=107) | 78.9 (18.02) | 73.9 (21.06)
  Physical Change from Baseline (n=58, n=60) | -1.6 (18.27) | -3.5 (17.21)
  Emotional Baseline (n=107, n=107) | 67.2 (20.21) | 62.1 (23.29)
  Emotional Change from Baseline (n=58, n=60) | -1.7 (17.36) | 0.3 (20.10)
  Sociality Baseline (n=107, n=107) | 45.9 (22.09) | 46.1 (22.37)
  Sociality Change from Baseline (n=58, n=60) | 1.6 (12.26) | 1.6 (17.05)
  Face Scale Baseline (n=107, n=107) | 59.3 (20.75) | 59.3 (25.12)
  Face Scale Change from Baseline (n=58, n=60) | -1.3 (20.64) | -2.1 (21.73)

5. Secondary Outcome: Change From Baseline to 3 Months in Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) Lung Cancer Subscale (LCS)
Description: FACT-L LCS measured health-related quality of life (HR-QL) related to additional concerns of lung cancer. Original LCS subscale scores range from 0 to 28, but the scores were converted to scores with a range of 0 to 100 in this study. Higher scores represent better HR-QL.
Time Frame: Baseline (pre-dose), 3 Months after first dose of Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Number analyzed (Participants) | 108 | 108
units on a scale
  Baseline (n=107, n=107) | 71.5 (18.81) | 69.6 (18.52)
  Change from Baseline (n=58, n=60) | 3.0 (16.13) | 0.4 (18.63)

ADVERSE EVENTS:
Arm/Group | Pemetrexed 500 mg/m2 | Pemetrexed 1000 mg/m2
Serious Adverse Events (participants affected / at risk) | 19/114 | 21/111
Other Adverse Events (participants affected / at risk) | 114/114 | 111/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500 mg/m2 (N=114) | Pemetrexed 1000 mg/m2 (N=111)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 5 (8)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500 mg/m2 (N=114) | Pemetrexed 1000 mg/m2 (N=111)
Abdominal discomfort (Gastrointestinal disorders) | 6 (9) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 10 (12)
Constipation (Gastrointestinal disorders) | 28 (33) | 21 (31)
Diarrhoea (Gastrointestinal disorders) | 16 (23) | 15 (19)
Nausea (Gastrointestinal disorders) | 64 (187) | 64 (133)
Stomatitis (Gastrointestinal disorders) | 9 (12) | 13 (23)
Vomiting (Gastrointestinal disorders) | 33 (122) | 36 (54)
Chest pain (General disorders) | 6 (7) | 3 (10)
Face oedema (General disorders) | 6 (6) | 4 (5)
Fatigue (General disorders) | 18 (35) | 18 (25)
Feeling hot (General disorders) | 9 (13) | 12 (16)
Malaise (General disorders) | 46 (100) | 49 (92)
Oedema (General disorders) | 6 (11) | 10 (11)
Oedema peripheral (General disorders) | 7 (8) | 6 (7)
Pyrexia (General disorders) | 35 (62) | 49 (97)
Nasopharyngitis (Infections and infestations) | 14 (18) | 14 (19)
Alanine aminotransferase increased (Investigations) | 81 (227) | 82 (185)
Aspartate aminotransferase increased (Investigations) | 88 (271) | 88 (254)
Blood albumin decreased (Investigations) | 25 (53) | 44 (85)
Blood alkaline phosphatase increased (Investigations) | 35 (51) | 35 (64)
Blood bilirubin increased (Investigations) | 11 (22) | 19 (43)
Blood chloride decreased (Investigations) | 7 (11) | 5 (10)
Blood creatinine increased (Investigations) | 11 (15) | 13 (25)
Blood glucose increased (Investigations) | 22 (36) | 19 (42)
Blood lactate dehydrogenase increased (Investigations) | 71 (182) | 71 (130)
Blood potassium decreased (Investigations) | 3 (7) | 6 (18)
Blood potassium increased (Investigations) | 4 (4) | 7 (15)
Blood pressure increased (Investigations) | 4 (8) | 8 (12)
Blood sodium decreased (Investigations) | 10 (11) | 10 (16)
Blood urea increased (Investigations) | 12 (18) | 9 (22)
Blood urine present (Investigations) | 20 (26) | 13 (27)
C-reactive protein increased (Investigations) | 31 (96) | 41 (102)
Gamma-glutamyltransferase increased (Investigations) | 10 (11) | 11 (16)
Glucose urine present (Investigations) | 11 (20) | 8 (21)
Haemoglobin decreased (Investigations) | 59 (133) | 68 (152)
Lymphocyte count decreased (Investigations) | 56 (109) | 64 (163)
Neutrophil count decreased (Investigations) | 73 (280) | 74 (256)
Neutrophil count increased (Investigations) | 22 (38) | 37 (84)
Platelet count decreased (Investigations) | 54 (170) | 51 (145)
Platelet count increased (Investigations) | 15 (52) | 12 (43)
Protein total decreased (Investigations) | 12 (22) | 20 (28)
Protein urine present (Investigations) | 18 (27) | 16 (27)
Red blood cell count decreased (Investigations) | 46 (109) | 45 (82)
Urobilin urine present (Investigations) | 5 (5) | 6 (9)
Weight decreased (Investigations) | 20 (20) | 30 (34)
White blood cell count decreased (Investigations) | 80 (287) | 81 (274)
White blood cell count increased (Investigations) | 27 (49) | 37 (83)
Anorexia (Metabolism and nutrition disorders) | 56 (149) | 76 (157)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 10 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (17) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (24) | 15 (15)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (11) | 11 (24)
Dizziness (Nervous system disorders) | 8 (12) | 8 (9)
Dysgeusia (Nervous system disorders) | 4 (7) | 7 (12)
Headache (Nervous system disorders) | 16 (24) | 18 (29)
Hypoaesthesia (Nervous system disorders) | 8 (8) | 5 (6)
Insomnia (Psychiatric disorders) | 12 (13) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 16 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 13 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 7 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 8 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (13)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (19) | 13 (25)
Rash (Skin and subcutaneous tissue disorders) | 79 (128) | 87 (134)
Hot flush (Vascular disorders) | 5 (6) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days